CLINICAL TRIAL: NCT06336551
Title: Efficacy of Acceptance and Commitment Therapy as a Stand-Alone Treatment for Insomnia: Protocol of a Randomized Waitlist Controlled Trial
Brief Title: Acceptance and Commitment Therapy for Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Mathilde Looman, Clinical Psychology PhD student, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityAmsterdam
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Insomnia
Keywords: Acceptance and Commitment Therapy; ACT-I; stand-alone; efficacy; mechanisms; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy for insomnia (ACT-I) (Experimental): In this condition, participants receive five individual face-to-face 60-minute sessions of ACT-I psychotherapy within a 7-week treatment period.
  Interventions: Behavioral: Acceptance and Commitment Therapy for insomnia (ACT-I)
- Waitlist control (No Intervention): In this condition, participants fill out assessments only during a 7-week waiting period. After completing the post-assessment, participants in the control condition receive ACT-I treatment as well.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for insomnia (ACT-I) — During ACT-I patients are encouraged to let go of the struggle to control sleep and to focus on meaningful daytime activities. Treatment goals are addressed through ACT processes of creative hopelessness and self-as-context (session 1), acceptance (session 2), defusion (session 3), followed by values, committed action, and present moment awareness (sessions 4 and 5).
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy for insomnia (ACT-I)

SUMMARY:
Insomnia is a common sleep problem that impacts both physical and mental health. Acceptance and Commitment Therapy for Insomnia (ACT-I) is proposed as a promising new treatment for insomnia. However, its effectiveness without overlapping behavioral components of the current standard treatment, cognitive behavioral therapy, remains largely unknown.

The main goal of this clinical trial is to test the efficacy of stand-alone ACT-I in adults with insomnia, compared to a waitlist control group. The second goal is to explore the potential working mechanisms of ACT-I, using network intervention analysis.

Adults with insomnia will be randomized to an ACT-I or waitlist group. Both the ACT-I treatment and waiting period span 7 weeks. Assessments take place at baseline (pre), after 4 weeks (mid), and after 8 weeks (post), followed by a 3- and 6-month follow-up for the ACT-I group.

The main questions this RCT aims to answer are:

* Is ACT-I superior to a waitlist control group in improving insomnia severity (primary outcome) in addition to sleep diary measures, anxiety, depression, general mental health, and sleep-related quality of life (secondary outcomes)?
* How do networks of insomnia symptoms or potential treatment processes (i.e., psychological (in)flexibility, sleep-related arousal, dysfunctional cognitions, and sleep-related safety behaviors) develop during and following ACT-I?

ELIGIBILITY:
Inclusion Criteria:

* insomnia severity index score ≥ 15
* clinical insomnia disorder diagnosis, as confirmed by the SCID-S-5 insomnia interview
* age of 18 years or above
* proficiency in Dutch
* ability to come on-site for the treatment sessions

Exclusion Criteria:

* previously received ACT
* started psychotherapy within the last 6 months or currently awaiting psychotherapy
* changed psychoactive medication in the last 3 months
* diagnosis of psychosis or schizophrenia
* severe depressive complaints (BDI-II score ≥ 29) or active suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | Change from baseline to 8-weeks post-randomization
  Insomnia severity is assessed with the Insomnia Severity Index (ISI). The ISI consists of seven items evaluating insomnia symptoms on a 5-point scale (range: 0-28). Higher scores indicate greater severity of insomnia symptoms.

SECONDARY OUTCOMES:
Insomnia severity | Change from baseline to 4-weeks post-randomization
  Insomnia severity is assessed with the Insomnia Severity Index (ISI). The ISI consists of seven items evaluating insomnia symptoms on a 5-point scale (range: 0-28). Higher scores indicate greater severity of insomnia symptoms.
Insomnia severity | Change from baseline to 3-month follow-up (ACT-I group only)
  Insomnia severity is assessed with the Insomnia Severity Index (ISI). The ISI consists of seven items evaluating insomnia symptoms on a 5-point scale (range: 0-28). Higher scores indicate greater severity of insomnia symptoms.
Insomnia severity | Change from baseline to 6-month follow-up (ACT-I group only)
  Insomnia severity is assessed with the Insomnia Severity Index (ISI). The ISI consists of seven items evaluating insomnia symptoms on a 5-point scale (range: 0-28). Higher scores indicate greater severity of insomnia symptoms.
General well-being | Change from baseline to 4-weeks post-randomization
  General well-being is assessed with the Mental Health Continuum Short Form (MHC-SF), which includes 14 items rated on a 6-point scale (range: 0-70). Higher scores indicate greater well-being.
General well-being | Change from baseline to 8-weeks post-randomization
  General well-being is assessed with the Mental Health Continuum Short Form (MHC-SF), which includes 14 items rated on a 6-point scale (range: 0-70). Higher scores indicate greater well-being.
General well-being | Change from baseline to 3-month follow-up (ACT-I group only)
  General well-being is assessed with the Mental Health Continuum Short Form (MHC-SF), which includes 14 items rated on a 6-point scale (range: 0-70). Higher scores indicate greater well-being.
General well-being | Change from baseline to 6-month follow-up (ACT-I group only)
  General well-being is assessed with the Mental Health Continuum Short Form (MHC-SF), which includes 14 items rated on a 6-point scale (range: 0-70). Higher scores indicate greater well-being.
Sleep-related quality of life | Change from baseline to 4-weeks post-randomization
  Sleep-related quality of life is evaluated using the Glasgow Sleep Impact Index (GSII). Respondents define and rate their three main domains of sleep-related impairment on a Visual Analog Scale (range: 0-100). Higher scores indicate more sleep-related impairment.
Sleep-related quality of life | Change from baseline to 8-weeks post-randomization
  Sleep-related quality of life is evaluated using the Glasgow Sleep Impact Index (GSII). Respondents define and rate their three main domains of sleep-related impairment on a Visual Analog Scale (range: 0-100). Higher scores indicate more sleep-related impairment.
Sleep-related quality of life | Change from baseline to 3-month follow-up (ACT-I group only)
  Sleep-related quality of life is evaluated using the Glasgow Sleep Impact Index (GSII). Respondents define and rate their three main domains of sleep-related impairment on a Visual Analog Scale (range: 0-100). Higher scores indicate more sleep-related impairment.
Sleep-related quality of life | Change from baseline to 6-month follow-up (ACT-I group only)
  Sleep-related quality of life is evaluated using the Glasgow Sleep Impact Index (GSII). Respondents define and rate their three main domains of sleep-related impairment on a Visual Analog Scale (range: 0-100). Higher scores indicate more sleep-related impairment.
Anxiety symptoms | Change from baseline to 4-weeks post-randomization
  Anxiety symptoms are assessed with the Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A), featuring seven items rated on a 4-point scale (range: 0-21). Higher scores indicate more anxiety symptoms.
Anxiety symptoms | Change from baseline to 8-weeks post-randomization
  Anxiety symptoms are assessed with the Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A), featuring seven items rated on a 4-point scale (range: 0-21). Higher scores indicate more anxiety symptoms.
Anxiety symptoms | Change from baseline to 3-month follow-up (ACT-I group only)
  Anxiety symptoms are assessed with the Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A), featuring seven items rated on a 4-point scale (range: 0-21). Higher scores indicate more anxiety symptoms.
Anxiety symptoms | Change from baseline to 6-month follow-up (ACT-I group only)
  Anxiety symptoms are assessed with the Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A), featuring seven items rated on a 4-point scale (range: 0-21). Higher scores indicate more anxiety symptoms.
Depression symptoms | Change from baseline to 4-weeks post-randomization
  Depression symptoms are assessed with the Patient Health Questionnaire depression scale (PHQ-9), a nine-item questionnaire scored on a 4-point scale (range: 0-36). Higher scores indicate more depression symptoms.
Depression symptoms | Change from baseline to 8-weeks post-randomization
  Depression symptoms are assessed with the Patient Health Questionnaire depression scale (PHQ-9), a nine-item questionnaire scored on a 4-point scale (range: 0-36). Higher scores indicate more depression symptoms.
Depression symptoms | Change from baseline to 3-month follow-up (ACT-I group only)
  Depression symptoms are assessed with the Patient Health Questionnaire depression scale (PHQ-9), a nine-item questionnaire scored on a 4-point scale (range: 0-36). Higher scores indicate more depression symptoms.
Depression symptoms | Change from baseline to 6-month follow-up (ACT-I group only)
  Depression symptoms are assessed with the Patient Health Questionnaire depression scale (PHQ-9), a nine-item questionnaire scored on a 4-point scale (range: 0-36). Higher scores indicate more depression symptoms.
Sleep diary: total sleep time | Change from baseline to 4-weeks post-randomization
  Total sleep time (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate higher total sleep time.
Sleep diary: total sleep time | Change from baseline to 8-weeks post-randomization
  Total sleep time (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate higher total sleep time.
Sleep diary: total sleep time | Change from baseline to 3-month follow-up (ACT-I group only)
  Total sleep time (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate higher total sleep time.
Sleep diary: total sleep time | Change from baseline to 6-month follow-up (ACT-I group only)
  Total sleep time (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate higher total sleep time.
Sleep diary: sleep onset latency | Change from baseline to 4-weeks post-randomization
  Sleep onset latency (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer sleep onset latency.
Sleep diary: sleep onset latency | Change from baseline to 8-weeks post-randomization
  Sleep onset latency (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer sleep onset latency.
Sleep diary: sleep onset latency | Change from baseline to 3-month follow-up (ACT-I group only)
  Sleep onset latency (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer sleep onset latency.
Sleep diary: sleep onset latency | Change from baseline to 6-month follow-up (ACT-I group only)
  Sleep onset latency (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer sleep onset latency.
Sleep diary: wake after sleep onset | Change from baseline to 4-weeks post-randomization
  Wake after sleep onset (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer wake time after sleep onset.
Sleep diary: wake after sleep onset | Change from baseline to 8-weeks post-randomization
  Wake after sleep onset (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer wake time after sleep onset.
Sleep diary: wake after sleep onset | Change from baseline to 3-month follow-up (ACT-I group only)
  Wake after sleep onset (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer wake time after sleep onset.
Sleep diary: wake after sleep onset | Change from baseline to 6-month follow-up (ACT-I group only)
  Wake after sleep onset (in minutes) is assessed with the consensus sleep diary (CSD). Higher scores indicate longer wake time after sleep onset.
Sleep diary: sleep efficiency | Change from baseline to 4-weeks post-randomization
  Sleep efficiency (in percentage) is assessed with the consensus sleep diary (CSD), calculated as the total sleep time*100 divided by the time in bed. Higher scores indicate higher sleep efficiency.
Sleep diary: sleep efficiency | Change from baseline to 8-weeks post-randomization
  Sleep efficiency (in percentage) is assessed with the consensus sleep diary (CSD), calculated as the total sleep time*100 divided by the time in bed. Higher scores indicate higher sleep efficiency.
Sleep diary: sleep efficiency | Change from baseline to 3-month follow-up (ACT-I group only)
  Sleep efficiency (in percentage) is assessed with the consensus sleep diary (CSD), calculated as the total sleep time*100 divided by the time in bed. Higher scores indicate higher sleep efficiency.
Sleep diary: sleep efficiency | Change from baseline to 6-month follow-up (ACT-I group only)
  Sleep efficiency (in percentage) is assessed with the consensus sleep diary (CSD), calculated as the total sleep time*100 divided by the time in bed. Higher scores indicate higher sleep efficiency.
Psychological flexibility | Change from baseline to 4-weeks post-randomization
  Psychological flexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological flexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological flexibility.
Psychological flexibility | Change from baseline to 8-weeks post-randomization
  Psychological flexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological flexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological flexibility.
Psychological flexibility | Change from baseline to 3-month follow-up (ACT-I group only)
  Psychological flexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological flexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological flexibility.
Psychological flexibility | Change from baseline to 6-month follow-up (ACT-I group only)
  Psychological flexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological flexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological flexibility.
Psychological inflexibility | Change from baseline to 4-weeks post-randomization
  Psychological inflexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological inflexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological inflexibility.
Psychological inflexibility | Change from baseline to 8-weeks post-randomization
  Psychological inflexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological inflexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological inflexibility.
Psychological inflexibility | Change from baseline to 3-month follow-up (ACT-I group only)
  Psychological inflexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological inflexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological inflexibility.
Psychological inflexibility | Change from baseline to 6-month follow-up (ACT-I group only)
  Psychological inflexibility is assessed with the Multidimensional Psychological Flexibility Inventory short form (MPFI-24). The subscale psychological inflexibility consists of 12 items, scored on a 6-point scale (range: 12-72). Higher scores indicate greater psychological inflexibility.
Sleep-related arousal | Change from baseline to 4-weeks post-randomization
  Sleep-related arousal will be assessed with the Pre-Sleep Arousal Scale (PSAS), which comprises 16 items scored on a 5-point scale (range: 16-80). Higher scores indicate higher sleep-related arousal.
Sleep-related arousal | Change from baseline to 8-weeks post-randomization
  Sleep-related arousal will be assessed with the Pre-Sleep Arousal Scale (PSAS), which comprises 16 items scored on a 5-point scale (range: 16-80). Higher scores indicate higher sleep-related arousal.
Sleep-related arousal | Change from baseline to 3-month follow-up (ACT-I group only)
  Sleep-related arousal will be assessed with the Pre-Sleep Arousal Scale (PSAS), which comprises 16 items scored on a 5-point scale (range: 16-80). Higher scores indicate higher sleep-related arousal.
Sleep-related arousal | Change from baseline to 6-month follow-up (ACT-I group only)
  Sleep-related arousal will be assessed with the Pre-Sleep Arousal Scale (PSAS), which comprises 16 items scored on a 5-point scale (range: 16-80). Higher scores indicate higher sleep-related arousal.
Dysfunctional sleep-related cognitions | Change from baseline to 4-weeks post-randomization
  Dysfunctional sleep-related cognitions will be evaluated by the short form of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16), which includes 16 items scored on an 11-point agreement scale (range: 0-160). Higher scores indicate more dysfunctional sleep-related cognitions.
Dysfunctional sleep-related cognitions | Change from baseline to 8-weeks post-randomization
  Dysfunctional sleep-related cognitions will be evaluated by the short form of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16), which includes 16 items scored on an 11-point agreement scale (range: 0-160). Higher scores indicate more dysfunctional sleep-related cognitions.
Dysfunctional sleep-related cognitions | Change from baseline to 3-month follow-up (ACT-I group only)
  Dysfunctional sleep-related cognitions will be evaluated by the short form of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16), which includes 16 items scored on an 11-point agreement scale (range: 0-160). Higher scores indicate more dysfunctional sleep-related cognitions.
Dysfunctional sleep-related cognitions | Change from baseline to 6-month follow-up (ACT-I group only)
  Dysfunctional sleep-related cognitions will be evaluated by the short form of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16), which includes 16 items scored on an 11-point agreement scale (range: 0-160). Higher scores indicate more dysfunctional sleep-related cognitions.
Sleep-related safety behaviors | Change from baseline to 4-weeks post-randomization
  Sleep-related safety behaviors will be measured with the sleep-related behaviors questionnaire short form (SRBQ-20), which consists of 20 items on coping with fatigue or improving sleep, scored on a 5-point scale (range: 0-80), with higher scores indicating more sleep-related safety behavior.
Sleep-related safety behaviors | Change from baseline to 8-weeks post-randomization
  Sleep-related safety behaviors will be measured with the sleep-related behaviors questionnaire short form (SRBQ-20), which consists of 20 items on coping with fatigue or improving sleep, scored on a 5-point scale (range: 0-80), with higher scores indicating more sleep-related safety behavior.
Sleep-related safety behaviors | Change from baseline to 3-month follow-up (ACT-I group only)
  Sleep-related safety behaviors will be measured with the sleep-related behaviors questionnaire short form (SRBQ-20), which consists of 20 items on coping with fatigue or improving sleep, scored on a 5-point scale (range: 0-80), with higher scores indicating more sleep-related safety behavior.
Sleep-related safety behaviors | Change from baseline to 6-month follow-up (ACT-I group only)
  Sleep-related safety behaviors will be measured with the sleep-related behaviors questionnaire short form (SRBQ-20), which consists of 20 items on coping with fatigue or improving sleep, scored on a 5-point scale (range: 0-80), with higher scores indicating more sleep-related safety behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Looman I Mathilde, MSc, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon requests.